CLINICAL TRIAL: NCT06315400
Title: Double-blind, Multicenter, Randomized, Placebo-controlled Study to Investigate the Efficacy, Safety and Tolerability of Ingavirin®, 60 mg Capsules in the Treatment of Influenza and Other Acute Respiratory Viral Infections in Children Aged 13-17 Years.
Brief Title: Efficacy and Safety of Ingavirin®, Capsules, 60 mg, in Children With Influenza and Other Acute Respiratory Viral Infections
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ING-07-2023
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-02

CONDITIONS: Influenza, Human; Acute Respiratory Infection; Common Cold
MeSH Terms: conditions — Influenza, Human; Common Cold | interventions — pentanedioic acid imidazolyl ethanamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ingavirin®, capsules, 60 mg (Experimental): Ingavirin® will be administered once a day (60 mg/day) for 5 days on top of standard therapy.
  Interventions: Drug: Ingavirin®
- Placebo (Placebo Comparator): Placebo will be administered once a day for 5 days on top of standard therapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ingavirin® — 60 mg/day for 5 days
  Arms: Ingavirin®, capsules, 60 mg
Drug: Placebo — 1 capsule/day for 5 days
  Arms: Placebo

SUMMARY:
The study is planned to evaluate the therapeutic efficacy and safety of Ingavirin®, capsules, 60 mg, in the treatment of influenza or other acute respiratory infections in children from 13 to 17 years compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 13 to 17 years inclusive.
2. Clinically established diagnosis of influenza or acute respiratory viral infection based on the presence of body temperature > 37.5 °C and at least 1 of the following symptoms of intoxication syndrome, and at least 1 manifestation of catarrhal syndrome: symptoms of intoxication syndrome (headache, chills, weakness, brokenness, eyeball pain, nausea); catarrhal syndrome (sore throat, rhinitis, pharyngitis, laryngitis, cough).
3. Laboratory-confirmed diagnosis of influenza or acute respiratory viral infections using one or more of the following viral antigen detection methods.
4. Uncomplicated course of influenza or ARVI.
5. Interval between the onset of the first symptoms of the disease and inclusion in the study no more than 36 h.
6. Availability of an informed consent form signed by one of the parents (or legal representatives) of the child for participation in the study.
7. For patients 14 years and older, a signed informed consent form for participation in the study.

Exclusion Criteria:

1. Hypersensitivity to any of the components included in the Ingavirin®.
2. Complicated course of influenza and acute respiratory viral infections (clinically and laboratory determined bacterial infection).
3. Taking antiviral drugs (antiviral agents, interferons, interferon inducers and drugs with immunomodulatory effect) or systemic antibacterial agents 7 days prior to the Screening Visit.
4. Severe influenza with signs of cardiovascular failure and other manifestations of infectious-toxic shock, as well as with the presence of neuroinfection syndrome (encephalic and meningoencephalic reactions).
5. Signs of viral pneumonia (presence of two or more of the following symptoms: dyspnea, chest pain when coughing, systemic cyanosis, dulling of the percussion sound with symmetric evaluation of the upper and lower lungs).
6. Infectious diseases suffered during the last week before inclusion of the patient in the study.
7. "Frequently ill children" (frequency of acute respiratory illnesses during the last year 6 times or more).
8. A history of bronchial asthma.
9. A history of increased seizure activity.
10. Severe, decompensated or unstable somatic diseases (any diseases or conditions that threaten the patient's life or worsen the patient's prognosis, as well as make it impossible to conduct a clinical trial in the patient).
11. History of oncologic diseases, HIV infection, tuberculosis.
12. Diabetes mellitus, lactose intolerance, lactase deficiency, glucose-galactose malabsorption, sucrose/isomaltase deficiency, fructose intolerance, hereditary disorders of glucose absorption, glucose-6-phosphate dehydrogenase deficiency.
13. Participation in a clinical drug trial less than 3 months prior to the start of the study.
14. Immunization of the patient 14 days prior to the Screening Visit.
15. The need for concomitant therapy with any of the drugs listed under "Prohibited Concomitant Treatment".
16. Any other concomitant somatic diseases or conditions that, in the opinion of the investigator, make it difficult to interpret the results of treatment or result in the inability to perform the procedures in this clinical trial or pose a risk to the patient in participating in the study.
17. For female patients, a positive urine pregnancy test if menstrual cycle is present.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with normalization of body temperature at Visit 3 (Day 3) | Day 0 - Day 21±1
  Percentage of patients with body temperature <37ºС with no rise above these values in the subsequent period until Visit 7

SECONDARY OUTCOMES:
Timeframe for normalization of body temperature from the start of treatment, measured in hours | Day 0 - Day 21±1
  Time (hours) to reach body temperature <37ºС with no rise above these values in the subsequent period until Visit 7 (Day 21±1)
Time of cough disappearance from the moment of treatment initiation | Day 0 - Day 21±1
  Disappearance of cough; no recurrence of cough in the following days of observation
Percentage of patients with absence of catarrhal syndrome | Day 0 - Day 21±1
  Percentage of patients with disappearance of all manifestations; no recurrence on subsequent days of follow-up) at Visit 3 (Day 3)
Percentage of patients with absence of intoxication syndrome | Day 0 - Day 21±1
  Percentage of patients with disappearance of all manifestations; no recurrence on subsequent days of follow-up) at Visit 3 (Day 3)
Average body temperature on days 1, 2, 3, 4 and 5 from the start of therapy | Day 1 - Day 5
  Average body temperature (two measurements per a day)
Percentage of patients with complications of influenza/acute respiratory infection that developed between days 1-6 and days 1-21 from the start of study drug administration | Day 0 - Day 21±1
  Percentage of patients with at least one complication of disease
Percentage of patients with severe complications of influenza/acute respiratory infection that developed between days 1-6 and days 1-21 from the start of study drug administration | Day 0 - Day 21±1
  Percentage of patients with at least one severe complication of disease
Assessment of vital signs: blood pressure | Day 1, Day 3, Day 6
  Blood pressure, mmHg
Assessment of vital signs: heart rate | Day 1, Day 3, Day 6
  Heart rate, bpm
Assessment of vital signs: respiratory rate | Day 1, Day 3, Day 6
  Respiratory rate, bpm
Assessment of vital signs: body temperature | Day 1 - Day 6
  Temperature, ºС
Evaluation of concomitant therapy | Day 0 - Day 21±1
  Number and types of concomitant therapy
Laboratory evaluation: leukocyte formula | Day 1, Day 6
  Precentage of white blood cells of different types
Laboratory evaluation: hemoglobin | Day 1, Day 6
  Hemoglobin, g/L
Laboratory evaluation: leukocyte count | Day 1, Day 6
  Cell/mL
Laboratory evaluation: platelet count | Day 1, Day 6
  Cell/mL
Laboratory evaluation: red blood cell count | Day 1, Day 6
  Cell/mL
Laboratory evaluation: hematocrit | Day 1, Day 6
  Hematocrit, %
Laboratory evaluation: erythrocyte sedimentation rate | Day 1, Day 6
  mm/h
Laboratory evaluation: blood glucose | Day 1, Day 6
  mmol/L
Laboratory evaluation: total protein | Day 1, Day 6
  g/L
Laboratory evaluation: total bilirubin | Day 1, Day 6
  mcmol/L
Laboratory evaluation: AST | Day 1, Day 6
  U/L
Laboratory evaluation: ALT | Day 1, Day 6
  U/L
Laboratory evaluation: creatinine | Day 1, Day 6
  mcmol/L
Laboratory evaluation: urea | Day 1, Day 6
  mmol/L
Laboratory evaluation: triglycerides | Day 1, Day 6
  mmol/L
Laboratory evaluation: urinalysis | Day 1, Day 6
  Urune color, transparency, specific gravity, pH, presence of protein, glucose, bilirubin, microscopy of urine sediment (epithelium, erythrocytes, leukocytes, cylinders, bacteria, salts)
Frequency of adverse events (AEs) and serious adverse events (SAEs) | Day 0 - Day 21±1
  Total number and frequency of AEs and SAEs stratified by severity and frequency
Percentage of patients who discontinued study due to AE/SAE | Day 0 - Day 21±1
  Percentage of patients who discontinued study participation early due to the occurrence of AE/SAE and time to dropout due to AE/SAE

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - GBOU VPO "Rostov State Medical University" of Ministry of Health of Russian Federation, Rostov-on-Don
  - GBOU VPO "Siberia State Medcial University" of Ministry of Health of Russian Federation, Tomsk
  - GBOU VPO "Yaroslavl State Medical University" of Ministry of Health of Russian Federation, Yaroslavl

IPD SHARING:
Plan to Share IPD: Undecided